CLINICAL TRIAL: NCT06924788
Title: Video-Conferenced Stress Management and Relaxation Training (VSMART) For Alabama Breast Cancer Survivors
Acronym: VSMART
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Chloe Taub, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300014220; UAB (Other: UAB)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breast cancer survivors receiving stress management program (Experimental): Breast cancer survivors receiving stress management program
  Interventions: Behavioral: Video-Conferenced Stress Management and Relaxation Training (VSMART)

INTERVENTIONS:
Behavioral: Video-Conferenced Stress Management and Relaxation Training (VSMART) — 10 week stress management group discussions

SUMMARY:
In a sample of Alabama breast cancer survivors, the proposed study tests the feasibility and acceptability of a stress management program that has been shown to improve health and wellbeing in a general population of patients with a history of breast cancer. The study will also get feedback (e.g., implementation barriers and facilitators) from relevant stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivor
* Currently living in Alabama
* Living in neighborhood with high deprivation index

Exclusion Criteria:

* Non-Alabama resident
* No history of breast cancer
* Living in neighborhood with low deprivation index

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of people enrolled out of contacted | At time of enrollment
  30% enrolled of contacted for feasibility threshold

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Taub, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No